CLINICAL TRIAL: NCT01760928
Title: Guidance of Patients With Asthma During Preparation and During Expedition to the Aconcagua Mountain
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dr. Lieven Dupont, Prof. dr., Universitaire Ziekenhuizen KU Leuven
Other Study IDs: ML9478
Record Dates: First submitted 2012-12-21; First posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — induced sputum cells and peripheral blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Asthma patients: all

SUMMARY:
A selection of asthma patients were followed during preparation to climb the Aconcagua mountain. The primary goal of this follow up was to optimize patients' asthma status. Also during expedition, these patients were daily consulted by a physician. All data obtained during preparation and expedition will now be retrospectively analyzed.

DETAILED DESCRIPTION:
Preparation phase:

Eighteen asthma patients were selected based on physical and medical characteristics. During the year of preparation, several time points of evaluation were planned: evaluation at baseline, maximal exercise test in hypoxia (FiO2: 11%), 24hour stay at cold air environment.

At baseline, medical history was evaluated and clinical examination, ECG, lung function, Fraction of exhaled NO measurement and histamine provocation were performed.

During a second visit, patients stayed for approximately one hour in a chamber to simulate high altitude (FiO2:11%) and performed a maximal exercise test after 30 minutes of rest. Oxygen saturation, ECG and oxygen consumption were continuously monitored. Lung function and fraction of exhaled NO were assessed before and after the test. Also, peripheral blood was drawn before and after the test. This test allowed us to identify whether patients may develop acute mountain sickness later on during expedition.

During a third visit, patients stayed for 24 hours in a indoor ski centre to practice climbing techniques, building up a tent and working with the specialized materials. Temperature at the ski piste varies between -5°C and -10°C. Lung function, fraction of exhaled NO and induced sputum was assessed before and after the stay at the ski centre.

During the expedition, clinical status, heart rate and oxygen saturation were measured daily. Also, lung function and fraction of exhaled NO were regularly measured. A screening for acute mountain sickness was performed daily. Asthmatics patients were supported by two pulmonologist. Before and after expedition, spirometry, histamine provocation and induced sputum were performed.

ELIGIBILITY:
Inclusion Criteria:

* asthma patient
* positive histamine provocation

Exclusion Criteria:

* exacerbation during the year prior to inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: asthmatics with well-controlled asthma
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To assess the type of airway inflammation evoked by exercise, hypoxia and cold air | one year
  Sputum cells and cytokine messenger ribonucleic acid will be analyzed to determine the type of airway inflammation that is induced by several triggers (exercise, hypoxia and cold air)

SECONDARY OUTCOMES:
To predict the occurrence of acute mountain sickness during an expedition to the Aconcagua mountain | one year
  * Mean Lake Louise Score in subjects
  * Number of subjects with Lake Louise Score > 5
  * Mean change in daily asthma symptom score
  * Mean change in Asthma control test score
  * Number of participants with an acute asthma exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Sven S Seys, MSc, Study Director — lab of clinical immunology, O&N I Herestraat 49 - bus 811, 3000 Leuven, België
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium